CLINICAL TRIAL: NCT05460377
Title: Assessing Immunogenicity of Intramuscular Sabin Inactivated Poliovirus Vaccine and Non-inferiority of Intradermal Fractional Inactivated Poliovirus Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); World Health Organization (Other); Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-21092
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Poliomyelitis
Keywords: Sabin Inactivated Poliovirus Vaccine; poliovirus vaccines; immunization; antibodies
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IMBCAMS Sabin IPV full dose at 14 weeks and 9 months (Active Comparator): Participants will receive two full doses of Sabin IPV intramuscularly at 14 weeks and 9 months produced by Institute of Medical Biology Chinese Academy of Medical Sciences, Kunming (IMBCAMS).
  Interventions: Biological: Full dose Sabin Inactivated Poliovirus Vaccine produced by IMBCAMS
- IMBCAMS Sabin IPV fractional dose at 14 weeks and 9 months (Active Comparator): Participants will receive two fractional (1/5) doses of Sabin IPV intradermally at 14 weeks and 9 months produced by Institute of Medical Biology Chinese Academy of Medical Sciences, Kunming (IMBCAMS).
  Interventions: Biological: Fractional (1/5) Dose Sabin Inactivated Poliovirus Vaccine produced by IMBCAMS
- BIBP Sabin IPV full dose at 14 weeks and 9 months (Active Comparator): Participants will receive two full doses of Sabin IPV intramuscularly at 14 weeks and 9 months produced by Beijing Bio Institute Biological Products (BIBP).
  Interventions: Biological: Full dose Sabin Inactivated Poliovirus Vaccine produced by BIBP
- BIBP Sabin IPV fractional dose at 14 weeks and 9 months (Active Comparator): Participants will receive two fractional (1/5) doses of Sabin IPV intradermally at 14 weeks and 9 months produced by Beijing Bio Institute Biological Products (BIBP).
  Interventions: Biological: Fractional (1/5) dose Sabin Inactivated Poliovirus Vaccine produced by BIBP

INTERVENTIONS:
Biological: Full dose Sabin Inactivated Poliovirus Vaccine produced by IMBCAMS — The Sabin antigen content is 30, 32 and 45 D-antigen units (DU) for types 1, 2 and 3, respectively and will be delivered intramuscularly by needle and syringe.
  Arms: IMBCAMS Sabin IPV full dose at 14 weeks and 9 months
Biological: Fractional (1/5) Dose Sabin Inactivated Poliovirus Vaccine produced by IMBCAMS — The Sabin antigen content is 30, 32 and 45 D-antigen units (DU) for types 1, 2 and 3, respectively and will be delivered intradermally by needle and syringe.
  Arms: IMBCAMS Sabin IPV fractional dose at 14 weeks and 9 months
Biological: Full dose Sabin Inactivated Poliovirus Vaccine produced by BIBP — The Sabin antigen content is 15 DU, 45 DU, 45 DU for types 1, 2, and 3, respectively and will be delivered intramuscularly by needle and syringe
  Arms: BIBP Sabin IPV full dose at 14 weeks and 9 months
Biological: Fractional (1/5) dose Sabin Inactivated Poliovirus Vaccine produced by BIBP — The Sabin antigen content is 15 DU, 45 DU, 45 DU for types 1, 2, and 3, respectively and will be delivered intradermally by needle and syringe
  Arms: BIBP Sabin IPV fractional dose at 14 weeks and 9 months

SUMMARY:
This is an open label and off label, phase IV, randomized clinical trial that will compare the immune response among infants that receive either two full doses of Sabin IPV intramuscularly or two fractional (1/5) dose of Sabin IPV intradermally at 14 weeks and 9 months of age from two different manufacturers.

DETAILED DESCRIPTION:
After OPV cessation, which is expected within a year of polio eradication certification, IPV will be the only polio vaccine used in essential immunization programs. SAGE has recommended a two-dose intramuscular IPV or intradermal fractional IPV (fIPV) schedule after OPV cessation. While it is expected that there shall be sufficient IPV available - in large part because of several manufacturers establishing production of IPV using Sabin strains (sIPV) - it is dependent on these manufacturers being able to meet promised product development and manufacturing timeline and meet WHO prequalification. It is likely that countries that have introduced intradermal fIPV pre-eradication will continue to use intradermal fIPV post-eradication. Therefore, it is important to generate evidence on immunogenicity of intradermal fractional sIPV in addition to intramuscular sIPV for the schedule recommended by SAGE.

This clinical trial assesses and compares the immunogenicity of full and fractional (1/5) dose Sabin IPV given at 14 weeks and 9 months of age from two different manufacturers. Healthy infants 6 weeks of age will be enrolled in Dhaka, Bangladesh, and randomized to one of four arms:

A. IMBCAMS full dose sIPV at 14 weeks and 9 months B. IMBCAMS fractional dose sIPV at 14 weeks and 9 months C. BIBP full dose sIPV at 14 weeks and 9 months D. BIBP fractional dose sIPV at 14 weeks and 9 months

Participants will be followed until 10 months of age through clinic visits. Blood samples will be collected for measuring immune response.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 6 weeks of age (range: 42-48 days).
* Parents that consent for participation in the full length of the study (i.e., 34 weeks).
* Parents that are able to understand and comply with planned study procedures.

Exclusion Criteria:

* A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member.
* A diagnosis or suspicion of bleeding disorder that would contraindicate parenteral administration of sIPV or collection of blood by venepuncture.
* Acute diarrhoea, infection or illness at the time of enrollment (6 weeks of age) that would require infant's admission to a hospital.
* Acute vomiting and intolerance to liquids within 24 hours before the enrollment visit (6 weeks of age).
* Evidence of a chronic medical condition identified by a study medical officer during physical exam.
* Receipt of any polio vaccine (OPV or IPV) before enrollment based upon documentation or parental recall.
* Known allergy/sensitivity or reaction to polio vaccine, or its contents.
* Infants from multiple births. Infants from multiple births will be excluded because the infant(s) who is/are not enrolled would likely receive OPV through routine immunization and transmit vaccine poliovirus to the enrolled infant.
* Infants from premature births (<37 weeks of gestation).

Ages: 42 Days to 48 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1224 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Vaccine response | Measured 4 weeks after administration of study vaccine
  Dichotomous (yes/no) variable defined as participants who are either seronegative (<1:8 titers) at baseline who become seropositive (≥1:8) after vaccination (seroconversion) or participants who demonstrate a four-fold rise in titers after vaccination between two specimens, e.g. a change from 1:8 to 1:32, after adjusting for expected decay in maternal antibodies. Antibody titers at 14 weeks of age will be the starting point for the expected decline in maternal antibodies, assuming at half-life of 28 days.

SECONDARY OUTCOMES:
Reciprocal antibody titers | Measured 4 weeks after administration of study Vaccine
  Variable of the observed reciprocal antibody titer results.
Priming | Measured 7 days after challenge dose (e.g. 9 months + 7 days)
  Dichotomous (yes/no) variable defined as participants who are either seronegative (<1:8 titers) at baseline who become seropositive (≥1:8) after vaccination (seroconversion) or participants who demonstrate a four-fold rise in titers after vaccination between two specimens, e.g. a change from 1:8 to 1:32, after adjusting for expected decay in maternal antibodies. Antibody titers at 14 weeks of age will be the starting point for the expected decline in maternal antibodies, assuming at half-life of 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Khalequ Zaman, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Icddr,B Study Clinics, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No